CLINICAL TRIAL: NCT00412464
Title: A Pilot Dose-finding and Pharmacokinetic Study of Fondaparinux in Children With Deep Vein Thrombosis or Heparin-induced Thrombocytopenia
Brief Title: Pilot Dose Finding and Pharmacokinetic Study of Fondaparinux in Children With Thrombosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Guy Young, Children's Hospital Los Angeles
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3091
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-10

CONDITIONS: Thrombosis; Heparin-induced Thrombocytopenia
Keywords: fondaparinux; thrombosis; heparin-induced thrombocytopenia; pediatrics
MeSH Terms: conditions — Thrombosis | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fondaparinux — Fondaparinux 0.1 mg/kg (up to 7.5 mg max initial dose) once daily for up to 21 days.
  Other Names: Arixtra

SUMMARY:
This study will evaluate the use of a blood thinner, fondaparinux, which is approved for use in adults (not in children) in a children aged 1-18 years. Subject with a blood clot (thrombosis) or heparin-induced thrombocytopenia who need to be on a blood thinner will be eligible to participate. Subjects will receive a once daily dose of fondaparinux followed by blood tests at 2, 4, 12, and 24 hours after the first dose in order to determine the proper dose for this age group. The hypothesis is that children receiving fondaparinux will be able to receive a once daily dose. The currently available alternative agent, enoxaparin, needs to be given twice daily. In addition, an evaluation of the safety of this medication will be made by assessing for side effects, especially bleeding.

DETAILED DESCRIPTION:
This clinical trial will assess the pharmacokinetics and safety of the novel anticoagulant, fondaparinux sodium (Arixtra) in pediatric patients with thromboembolism. Currently available anticoagulants have significant limitations especially as it applies to the pediatric population. Thus novel agents with improved pharmacologic properties are needed to improve the care of this increasingly recognized complication in children. Furthermore, the only available agent for long-term anticoagulation in children with heparin-induced thrombocytopenia is warfarin. Anticoagulation with warfarin in the pediatric population is problematic due to its narrow therapeutic index and the numerous drug and food interactions necessitating frequent laboratory monitoring. In addition, oral administration of warfarin (which cannot be compounded to a liquid) is difficult in young children. Thus a novel agent for this condition is needed and fondaparinux does not cross-react with heparin antibodies. The aims of the study are to determine the proper dosing regimen (dose and interval) and safety in patients less than 18 years of age with thrombosis or heparin-induced thrombocytopenia. Another aim is to assess the utility of thromboelastography as a monitoring tool for patients on fondaparinux. This will be a pilot study which will have a total of 24 patients in 3 age cohorts with 8 patients per cohort as follows: 1-5 years, 6 -12 years, and 12-18 years as the pharmacokinetics of medications differ by age. Patients will receive an initial dose of 0.1mg/kg subcutaneously daily. After the first dose, fondaparinux levels will be drawn at 2,4,12, and 24 hours after administration. Dose adjustments will be made based on the 4 hour (peak) level and trough levels at 12 and 24 hours will determine if daily dosing is feasible. Thromboelastography will be performed at 2 or 4 hours and 24 hours with the results correlated with the plasma activity level. Safety will be assessed by physical examination, laboratory testing, and if necessary diagnostic imaging to determine the incidence of minor and major bleeding. Pharmacokinetic analyses as well as safety and efficacy determinations will be made which will provide valuable information on this promising new anticoagulant for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 year and 18 years of age.
* The presence of documented venous or arterial thrombosis confirmed by diagnostic imaging.
* Weight greater than 8.3 kg.
* Signed informed consent/assent.

Exclusion Criteria:

* Patients with active bleeding.
* Patients with planned invasive procedures less than 2 weeks from the time of enrollment.
* Patients with a contraindication to anticoagulation.
* Patients receiving thrombolytic agents.
* Patients with an INR>1.5 or an activated partial thromboplastin time (PTT)>40 seconds.
* Patients with a creatinine level above 1.2 times the upper limit of normal expected for age.
* Children <1 year of age.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Young, MD, Principal Investigator — Children's Hospital of Orange County
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Result] Young G, Yee FL, Khanna R, O'Brien D, Nugent DJ. Fondaparinux for the Treatment of Thrombosis in Children: A Prospective, Dose-Finding, Pharmacodynamic and Safety Study. Blood (ASH Annual Meeting Abstracts), Nov 2009; 114: 3130.
- [Result] Young G, Yee DL, O'Brien SH, Khanna R, Barbour A, Nugent DJ. FondaKIDS: a prospective pharmacokinetic and safety study of fondaparinux in children between 1 and 18 years of age. Pediatr Blood Cancer. 2011 Dec 1;57(6):1049-54. doi: 10.1002/pbc.23011. Epub 2011 Feb 11. PMID 21319285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between September, 2006 and June, 2009 at 4 sites (Children's Hospital Los Angeles, Children's Hospital of Orange County, Texas Children's Hospital and Nationwide Children's Hospital). All subjects were in the inpatient units of these hospitals for the duration of their study participation.
Pre-assignment Details: All recruited subjects entered and completed the study.
Groups:
- Fondaparinux Group: Single arm group receiving fondaparinux 0.1 mg/kg.
Period: Overall Study
Arm/Group | Fondaparinux Group
Started | 24 (Age Groups: 1-5 Years (10); 6-12 Years (7); 13-18 years (7))
Completed | 24 (Age Groups: 1-5 Years (10); 6-12 Years (7); 13-18 years (7))
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Abnormal Lab Results Resulting in Adverse Events.
Description: The primary outcome measure was assessment of safety by reporting the number of abnormal lab results resulting in adverse events. Safety laboratory assessments are as follows: Liver and kidney toxicity will be determined by serial measurements of AST, ALT, total bilirubin, BUN and creatinine. Hematologic toxicity will be assessed by serial CBCs.
Time Frame: Study period which was up to 21 days of fondaparinux
Measure: Number; unit: Adverse Events
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
Adverse Events | 0

2. Primary Outcome: Therapeutic Plasma Concentration of Fondaparinux at 21 Days
Description: Subjects all had detailed pharmacokinetic measurements done which were subsequently analyzed in a population pharmacokinetic model. This model then informed the dosing recommendations that were published as a result of the study.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
mg/dL | 24 (0.001)

3. Primary Outcome: Bleeding Events
Description: Bleeding assessment Patients will be monitored for bleeding symptoms by physician and nursing assessment. Major bleeding will be defined as bleeding which is in a critical space (intracranial, retroperitoneal, or visceral) or leads to the need for blood transfusion. Minor bleeding will be all other bleeding and will be classified as clinically significant (i.e. If the physician has to take action to treat the minor bleed) or clinically insignificant (i.e. if the physician does not need to intervene to treat the minor bleed).
Time Frame: Study period which was up to 21 days of fondaparinux
Measure: Number; unit: Adverse Events
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
Adverse Events | 2

4. Primary Outcome: Adverse Events
Description: Adverse events will be defined as any untoward or unexpected event which can be a symptom, physical exam sign or laboratory abnormality. Adverse events will be classified as serious if they lead to prolonged hospitalization, re-hospitalization, transfer to an intensive care unit, or death. Adverse events will be categorized in terms of their likely association with fondaparinux as probably related, possibly related, unrelated, or unknown, and will be recorded according to standard adverse reporting guidelines for clinical trials.
Time Frame: Study period which was up to 21 days of fondaparinux
Measure: Number; unit: Adverse Events
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
Adverse Events | 0

5. Primary Outcome: Thrombocytopenic Events
Description: Patient's platelet counts should be kept above 50 x 10^9/L while on study with platelet transfusions as needed with the exception of patients enrolled under the HIT/ suspicion of HIT inclusion (platelet transfusions are contraindicated in HIT). With regards to study patients who experience progressive decreases in platelet count to below 50 x 10^9/L while receiving fondaparinux (excluding patients being treated for HIT or suspicion of HIT), fondaparinux will be discontinued.
Time Frame: Study period which was up to 21 days of fondaparinux
Measure: Number; unit: Adverse Events
Arm/Group | Fondaparinux Group
Number analyzed (Participants) | 24
Adverse Events | 0

ADVERSE EVENTS:
Arm/Group | Fondaparinux Group
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No